CLINICAL TRIAL: NCT05993702
Title: Single-arm, Multicentre Real-world Observational Study of TAS-102 in Combination With Regorafenib or Fruquintinib for Third-line and Above Advanced Colorectal Cancer
Brief Title: TAS-102 in Combination With Regorafenib or Fruquintinib for Third-line and Above Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Other Study IDs: PRAY
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: TAS 102; Regorafenib; Fruquintinib; Gastrointestinal Tumours
MeSH Terms: interventions — regorafenib; HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAS-102 in combination with regorafenib: (TAS102): Trifluridine tepipiridine tablets 35 mg/m2 twice a day, D1-5, D15-D19, 28 days as a cycle; (TKI: regorafenib: regorafenib capsules administered at a dose of 80 mg (2 tablets, each containing 40 mg regorafenib) once daily for a 28-day cycle)
  Interventions: Drug: regorafenib
- TAS-102 in combination with fruquintinib: TAS102: Trifluridine tepipiridine tablets 35 mg/m2 twice a day, D1-5, D15-D19, 28 days as a cycle; Fruquintinib: a dose of 3mg/dose administered orally once daily, continuously for 28 days as a cycle.
  Interventions: Drug: fruquintinib

INTERVENTIONS:
Drug: regorafenib — (TAS102): Trifluridine tepipiridine tablets 35 mg/m2 twice a day, D1-5, D15-D19, 28 days as a cycle; (TKI: regorafenib: regorafenib capsules administered at a dose of 80 mg (2 tablets, each containing 40 mg regorafenib) once daily for a 28-day cycle)
  Other Names: baiwange
  Groups: TAS-102 in combination with regorafenib
Drug: fruquintinib — TAS102: Trifluridine tepipiridine tablets 35 mg/m2 twice a day, D1-5, D15-D19, 28 days as a cycle; or Fruquintinib: a dose of 3mg/dose administered orally once daily, continuously for 28 days as a cycle.
  Other Names: elunate
  Groups: TAS-102 in combination with fruquintinib

SUMMARY:
This is a single-arm, multicentre real-world observational study of TAS-102 in combination with regorafenib or fruquintinib for third-line and above advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a single-arm, multicentre real-world observational study of TAS-102 in combination with regorafenib or fruquintinib for third-line and above advanced colorectal cancer.The purpose of the study is to evaluate the efficacy and safety of TAS-102 in combination with a regimen of regorafenib or fruquintinib for the treatment of advanced colorectal cancer in the third line and above.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18-75 years;
2. Patients with colorectal cancer diagnosed by histology or cytology;
3. Patients with metastatic colorectal cancer who have failed two or more standard therapies; patients are permitted to have received prior chemotherapy with fluorouracil, oxaliplatin, irinotecan, and other regimens, patients are permitted to receive EGFR and/or VEGF inhibitors, and patients are permitted to have received prior immunotherapy;
4. Have at least one measurable lesion according to the solid tumour efficacy evaluation criteria RECIST version 1.1; the measurable lesion should not have received local treatment such as radiotherapy (lesions located within the area of previous radiotherapy may also be selected as target lesions if progression is confirmed to have occurred and meets the RECIST 1.1 criteria);
5. ECOG PS score: 0 to 1; expected survival more than 3 months;
6. Oral medication is available;
7. have adequate organ and bone marrow function, i.e., meet the following criteria:

(1) Criteria for routine blood tests need to be met: Haemoglobin level (HB) ≥ 90 g/L (no transfusion within 28 days); Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelet count (PLT) ≥ 100×109/L. (2) Biochemical tests need to meet the following criteria: Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN) ; ALT and AST ≤ 2.5 ULN (ALT and AST ≤ 5 ULN if liver metastases are present); Cr ≤ 1.5 ULN or creatinine clearance (CCr) ≥ 60 ml/min; (Cockcroft-Gault formula) (3) Adequate coagulation function, defined as International Normalised Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN; 8) Pregnant or breastfeeding patients: 1) Females and males of childbearing potential must agree to use adequate contraception prior to entering the programme until at least 8 weeks after the last dose of study drug. The Investigator or designee is required to advise subjects on how to achieve adequate contraception. Appropriate contraception is defined in the study as any medically recommended method (or combination of methods) based on standard treatment 2) Women of childbearing age must have a negative serum or urine pregnancy test confirmed within 7 days prior to initiating treatment and must agree to record a negative result prior to entering the study.

Exclusion Criteria:

- study:

1. Patients with abnormal coagulation or a tendency to gastrointestinal bleeding on thrombolytic or anticoagulant medication, including active peptic ulcers with fecal occult blood++, vomiting blood or black stools within 3 months.
2. Prior or concurrent cancers with a primary site or histology different from CRC within the year of enrolment, with the exception of cured in situ cervical cancer, non-melanoma skin cancers, and superficial bladder tumours:staging Ta, Tis and T1 .
3. Arterial or venous thrombotic or embolic events, such as cerebrovascular accidents (including transient ischaemic attacks), deep vein thrombosis, or pulmonary embolism (except for appropriately treated catheter-associated venous thrombosis occurring more than 1 month after initiation of therapy), have occurred within 6 months prior to the start of treatment.
4. Major surgery, biopsy or significant traumatic injury within 28 days prior to the start of investigational therapy.
5. Unhealed wounds, ulcers, or fractures.
6. Patients with brain metastases and/or carcinomatous meningitis.
7. Congestive heart failure >New York Heart Association (NYHA) class 2.
8. Unstable angina (angina at rest), new onset angina (within the last 3 months). Myocardial infarction within 6 months prior to the start of treatment.
9. Arrhythmia requiring antiarrhythmic therapy (beta-blockers or digoxin permitted). Uncontrolled hypertension. (Systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical therapy).
10. Patients with pheochromocytoma
11. Pleural effusion or ascites causing respiratory restriction (≥ CTCAE grade 2 dyspnoea)
12. Active infection >NCI CTCAE2 level
13. interstitial lung disease with signs and symptoms at the time of informed consent
14. known hypersensitivity to any of the drugs in the study, to drugs of the same class as the study drug, or to excipients in dosage forms
15. use of CYP3A4 inhibitors or inducers
16. Participation in another clinical trial within 4 weeks prior to enrolment and receipt of the investigational drug and any concomitant therapy containing the investigational drug
17. have received radiotherapy within 4 weeks prior to enrolment and the lesion under observation in this study is in the target area of radiotherapy
18. Subjects with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within one year prior to screening
19. Subjects with comorbidities requiring long-term treatment with immunosuppressive drugs or systemic or topical corticosteroids at immunosuppressive doses (>10mg/day of prednisone or other equipotent hormones).
20. Received any anti-infective vaccine (e.g., influenza vaccine, varicella vaccine, neocoronavirus vaccine, etc.) within 4 weeks prior to enrolment.
21. Pregnancy or breastfeeding
22. Persistent proteinuria >3.5 g/24 hours by measurement of urine protein-creatinine ratio (grade 3, NCI-CTCAE version 5.0) in random urine samples.
23. Human immunodeficiency virus (HIV) positive
24. Hepatitis B virus surface antigen (HBsAg) positive and HBV DNA copy number positive (quantitative test ≥1000 cps/ml)
25. Positive blood test for chronic hepatitis C (HCV antibody positive)
26. renal failure requiring haemodialysis or peritoneal dialysis
27. Dehydration ≥ CTCAE Version 5.0 Level 1
28. Persons who are legally incompetent.
29. Any other clinically significant disease or condition that, in the opinion of the investigator, may affect adherence to the protocol, or the signing of the Informed Consent Form (ICF) by the subject, or make participation in this clinical trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients between the ages of 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | one year
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease Control Rate (DCR) | one year
  Determined using RECIST v1.1 criteria.
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | two years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — First Hospital of China Medical University

IPD SHARING:
Plan to Share IPD: No